CLINICAL TRIAL: NCT02574884
Title: Identification of Viral Variants Involved in the Transmission of Hepatitis C and Characterization of Antigenic and Functional Properties of Their Envelope Glycoproteins
Acronym: VINTAGE VHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AORT10-DB / VINTAGE VHC
Record Dates: First submitted 2015-10-02; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Recently infected subjects (Other): Actual population of blood donors primo-infected with HCV with specific intervention for the study : one blood sample during the inclusion visit
  Interventions: Procedure: Blood sample (act specific of blood withdrawal for the study)
- Retrospective cases (No Intervention): Population of infected blood donors in 2007, 2008 and 2009 No blood sample
- Individuals sources (Other): Specific intervention for the study : one blood sample during the inclusion visit
  Interventions: Procedure: Blood sample (act specific of blood withdrawal for the study)

INTERVENTIONS:
Procedure: Blood sample (act specific of blood withdrawal for the study) — Specific intervention : blood sample (3x7 ml in total)
  Arms: Individuals sources; Recently infected subjects

SUMMARY:
The study consists to Identify viral variants involved in the transmission of hepatitis C and characterize the antigenic and functional properties of their envelope glycoproteins at very early stage of infection (before seroconversion).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* agree to participate in this study (signing the consent form or information form signed and letter of no objection for subjects contaminated by blood exposure).

These criteria are specific to contaminated subjects:

* primary infection before development of HCV antibody (seroconversion): nucleic acid testing positive in the absence of HCV antibodies.

These criteria are specific to individual sources :

* HCV antibody positive.

Exclusion Criteria:

* refusal to participate
* private about freedom
* under guardianship
* under justice
* minor or major person unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
HCV serological markers | up to 30 months
  Immunoblot analysis from blood samples collected during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Chru de Tours, Tours, France, France